CLINICAL TRIAL: NCT00944034
Title: A Phase 2b, Open Label, Multi-Center, Extension Study to Evaluate the Safety, Tolerability and Immunogenicity of a Booster Dose of Novartis Meningococcal B Recombinant Vaccine Administered at 12, 18 or 24 Months of Age in Subjects Who Previously Received a Three-Dose Primary Series of the Novartis Meningococcal B Recombinant Vaccine as Infants in Study V72P12
Brief Title: Safety, Tolerability and Immunogenicity of Meningococcal B Recombinant Vaccine Administered as Booster Dose at 12, 18 or 24 Months of Age in Toddlers (12-24 Months) Primed With a Three-Dose Immunization Series as Infants in Study V72P12
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P12E1; 2009-011676-30
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal meningitis; prevention; vaccination; toddler
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal

ARMS (12):
- B+R246_12 (Experimental): Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age.
  Interventions: Biological: rMenB+OMV NZ with routine vaccinations
- B+R246_18 (Experimental): Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 18 months of age.
  Interventions: Biological: rMenB+OMV NZ with routine vaccinations
- B+R246_24 (Experimental): Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 24 months of age.
  Interventions: Biological: rMenB+OMV NZ with routine vaccinations
- B246_12 (Experimental): Previously received 3 doses of rMenB+OMV NZ vaccine at 2, 4 and 6 months of age and routine vaccines at 3, 5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age.
  Interventions: Biological: rMenB+OMV NZ
- B246_18 (Experimental): Previously received 3 doses of rMenB+OMV NZ vaccine at 2, 4 and 6 months of age and routine vaccines at 3,5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ at 18 months of age.
  Interventions: Biological: rMenB+OMV NZ
- B246_24 (Experimental): Previously received 3 doses of rMenB+OMV NZ vaccine at 2, 4 and 6 months of age and routine vaccines at 3, 5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ at 24 months of age.
  Interventions: Biological: rMenB+OMV NZ
- B+R234_12 (Experimental): Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ at 12 months of age.
  Interventions: Biological: rMenB+OMV NZ with routine vaccinations
- B+R234_18 (Experimental): Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 18 months of age.
  Interventions: Biological: rMenB+OMV NZ with routine vaccinations
- B+R234_24 (Experimental): Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 24 months of age.
  Interventions: Biological: rMenB+OMV NZ with routine vaccinations
- B12 14 (Experimental): Previously received two catch-up doses of rMenB+OMV NZ vaccine at 12 and14 months of age.
  Interventions: Biological: two doses of rMenB+OMV NZ
- B18 20 (Experimental): Previously received two catch-up doses of rMenB+OMV NZ vaccine at 18 and 20 months of age.
  Interventions: Biological: two doses of rMenB+OMV NZ
- B24 26 (Experimental): Previously received two catch-up doses of rMenB+OMV NZ vaccine at 24 and 26 months of age.
  Interventions: Biological: two doses of rMenB+OMV NZ

INTERVENTIONS:
Biological: rMenB+OMV NZ with routine vaccinations — rMenB+OMV NZ with routine vaccinations at 2, 4, and 6 months of age; random allocation in a 1:1:1 ratio to receive a booster dose of rMenB+OMV NZ at 12 months of age
  Arms: B+R246_12
Biological: rMenB+OMV NZ with routine vaccinations — rMenB+OMV NZ with routine vaccinations at 2, 4, and 6 months of age; random allocation in a 1:1:1 ratio to receive a booster dose of rMenB+OMV NZ at 18 months of age
  Arms: B+R246_18
Biological: rMenB+OMV NZ — rMenB+OMV NZ at 2, 4, and 6 months of age and routine vaccinations at 3, 5 and 7 months of age; random allocation in a 1:1:1 ratio to receive a booster dose of rMenB+OMV NZ at 12 months of age
  Arms: B246_12
Biological: rMenB+OMV NZ — rMenB+OMV NZ at 2, 4, and 6 months of age and routine vaccinations at 3, 5 and 7 months of age; random allocation in a 1:1:1 ratio to receive a booster dose of rMenB+OMV NZ at 18 months of age
  Arms: B246_18
Biological: rMenB+OMV NZ with routine vaccinations — rMenB+OMV NZ with routine vaccinations at 2, 3 and 4 months of age; random allocation in a 1:1:1 ratio to receive 1 booster dose of rMenB+OMV NZ at 12 months of age
  Arms: B+R234_12
Biological: rMenB+OMV NZ with routine vaccinations — rMenB+OMV NZ with routine vaccinations at 2, 3 and 4 months of age; random allocation in a 1:1:1 ratio to receive 1 booster dose of rMenB+OMV NZ at 18 months of age
  Arms: B+R234_18
Biological: two doses of rMenB+OMV NZ — two catch-up doses of rMenB+OMV NZ at 12 and 14 months of age.
  Arms: B12 14
Biological: rMenB+OMV NZ with routine vaccinations — rMenB+OMV NZ with routine vaccinations at 2, 4, and 6 months of age; random allocation in a 1:1:1 ratio to receive a booster dose of rMenB+OMV NZ at 24 months of age
  Arms: B+R246_24
Biological: two doses of rMenB+OMV NZ — two catch-up doses of rMenB+OMV NZ at 18 and 20 months of age
  Arms: B18 20
Biological: rMenB+OMV NZ — rMenB+OMV NZ at 2, 4, and 6 months of age and routine vaccinations at 3, 5 and 7 months of age; random allocation in a 1:1:1 ratio to receive a booster dose of rMenB+OMV NZ at 24 months of age
  Arms: B246_24
Biological: two doses of rMenB+OMV NZ — two catch-up doses of rMenB+OMV NZ at 24 and 26 months of age
  Arms: B24 26
Biological: rMenB+OMV NZ with routine vaccinations — rMenB+OMV NZ with routine vaccinations at 2, 3 and 4 months of age; random allocation in a 1:1:1 ratio to receive 1 booster dose of rMenB+OMV NZ at 12 (Group 3a), 18 (Group 3b) or 24 (Group 3c) months of age
  Arms: B+R234_24

SUMMARY:
This extension study V72P12E1 will investigate the safety, tolerability and immunogenicity of a fourth (booster) dose of rMenB+OMV NZ at 12, 18 and 24 months of age in subjects previously primed with rMenB+OMV NZ according to two different three-dose immunization schedules in infancy (2, 4 and 6 or 2, 3 and 4 months of age in the parent study V72P12). The study will also explore the bactericidal antibody persistence at 12, 18 and 24 months of age, following the two different immunization schedules, in order to identify the optimal timing for boosting. Two catch-up rMenB+OMV NZ doses will be given to unprimed, naïve toddlers at 12 (subjects enrolled in the control group of V72P12), 18 and 24 months of age (two new cohort of subjects enrolled). These subjects will generate data for assessing the safety and immunogenicity of a two-dose catch-up regimen at these ages, but will also serve as controls for a descriptive comparison of antibody persistence and booster responses for the other groups.

ELIGIBILITY:
Inclusion Criteria:

Follow-on participants of V72P12:

Healthy toddlers who completed Study V72P12, aged:

* 12 months or older - Groups 1a, 2a, 3a, 4
* 18 months (0/ +29 days window) - Groups 1b, 2b, 3b
* 24 months (0/ +29 days window) - Groups 1c, 2c, 3c

Naive subjects newly enrolled:

* Group 5: healthy 18-month-old toddlers (0/ +29 days window)
* Group 6: healthy 24-month-old toddlers (0/ +29 days window)

Exclusion Criteria:

* History of any meningococcal B vaccine administration (only for groups 5 and 6);
* Previous ascertained or suspected disease caused by N. meningitidis;
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component;
* Significant acute or chronic infection within the previous 7 days or axillary temperature major or equal to 38 degrees within the previous day
* Antibiotics within 6 days prior to enrollment;
* Any serious chronic or progressive disease;
* Known or suspected impairment or alteration of the immune system;
* Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1588 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- Belgium (7):
  - Avenue Albert 1er 185, 5000 Namur
  - Avenue Hippocrate 10, 1200 Brussels
  - Laarbeeklaan 101, 1090 Brussels
  - Lindendreef 1, 2020 Antwerpen
  - Sint Vincentiusstraat 20, 2018 Antwerpen
  - Stadsomvaart 11, 3500 Hasselt
  - Wilrijkstraat 10, 2650 Edegem
- Czechia (4):
  - Červený Kostelec
  - Kyjevska 44, 532 03 Pardubice
  - Ruskych Legii 352, 377 01 Jindrichuv Hradec
  - Trebesska 1575, 500 01 Hradec Kralove
- Germany (30):
  - Ahrensböker Str. 11, 23617 Stockelsdorf
  - Am Alten Hafen 117, 27568 Bremerhaven
  - Ammertalweg 7, 99086 Erfurt
  - Anne Frank Str.27, 75015 Bretten
  - Bucher Chaussee 1-3, 13125 Berlin
  - Christian-Bauer-Str.5, 73642 Welzheim
  - Deckertstr. 53, 33645 Bielefeld
  - Dingbängerweg 69, 48163 Münster
  - Elisenstr. 28, 63739 Aschaffenburg
  - Gartenstr. 3,76889 Schweigen
  - Großbottwarer Str. 47, 71720 Oberstenfeld
  - Hanseatenplatz 1, 25524 Itzehoe
  - Hauptstr. 165, 42579 Heiligenhaus
  - Hauptstr. 240, 77694 Kehl
  - Hauptstr. 46, 37083 Göttingen
  - Josef-Sugg-Str. 5, 88348 Bad Saulgau
  - Kapellenstraße 27, 47533 Kleve-Materborn
  - Kleinenbroicher Str. 68, 41352 Korschenbroich
  - Kuhtrift 8a, 34414 Warburg
  - Langenbeckstraße 1, 55101 Mainz
  - Lindenpromenade 34b, 39164 Wanzleben
  - Lindenstr. 9, 25524 Itzehoe
  - Marienstraße 2, 44866 Bochum
  - Maschstr. 8a, 49565 Bramsche
  - Mose-Stern-Str. 28, 41236 Mönchengladbach
  - Ostlandstr. 10, 32339 Espelkamp
  - Poststr. 10, 34225 Baunatal
  - Tangstedter Landstr 77, 22415 Hamburg
  - Wilhelmshöher Allee 109, 34121 Kassel
  - Würzburger Str. 1, 97941 Tauberbischofsheim
- Italy (10):
  - C.so Mazzini 18, 28100 Novar
  - Current Address: Via Luca Giordano N. 13, 50132 Firenze
  - Piazza Ospedale 10, 20900 Lodi
  - Via Commenda 9, 20122, Milano
  - Via Consolare Valeria 1, 98125 Messina
  - Via G.B.Grossi 74, 20157 Milano
  - Via Giustiniani,3, 35128 Padova
  - Via Pastore 1,16132 Genova
  - Via Siracusa, 45, 90143 Palermo
  - Viale Pieraccini N. 24 50139 Firenze
- Spain (16):
  - Avda. Rambleta, S/n Catarroja Valencia
  - C/ Tossal Del Rei Nº 7 Castellón de La Plana Castellón
  - Catarroja Esquina Ministro Serrano. Paiporta Valencia
  - Celestino Villamil, S/n Oviedo
  - Ctra. Anfondeguilla, S/n Vall Duixo Castellón
  - Isabel de Villena,2 Pabellón Valencia
  - Médico Fernando Moray de La Horra, 2 Acceso Y9 Valencia
  - Molí S/n Puçol Valencia
  - Pedro S/n Almazora Castellón
  - Pizarro, 22 Vigo Pontevedra
  - Plaza Blasco Ibañez, 4 Sagunto Valencia
  - Plaza Segovia S/n Valencia
  - República Argentina Nº 8, Valencia
  - Rosales, 23 La Eliana Valencia
  - Serreria,73 Valencia
  - Travesía Da Choupana, S/n Santiago de Compostela A Coruña
- United Kingdom (5):
  - University Hospitals Bristol, NHS Foundation Trust, Trust Headquarters, Marlborough Street, Bristol
  - South West Medicines for Children Research Network, Child Health Building, Royal Devon and Exeter NHS Foundation Trust, Barrack Road, Exeter
  - St. George's University of London, Cranmer Terrace, London
  - Oxford Vaccines Group, Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Old Road, Headington, Oxford
  - Centre for Clinical Vaccinology, Oxford

REFERENCES:
- [Derived] Bartolini E, Borgogni E, Bruttini M, Muzzi A, Giuliani M, Iozzi S, Petracca R, Martinelli M, Bonacci S, Marchi S, Brettoni C, Donati C, Torricelli G, Guidotti S, Domina M, Beninati C, Teti G, Felici F, Rappuoli R, Castellino F, Del Giudice G, Masignani V, Pizza M, Maione D. Immunological fingerprint of 4CMenB recombinant antigens via protein microarray reveals key immunosignatures correlating with bactericidal activity. Nat Commun. 2020 Oct 5;11(1):4994. doi: 10.1038/s41467-020-18791-0. PMID 33020485
- [Derived] Snape MD, Voysey M, Finn A, Bona G, Esposito S, Principi N, Diez-Domingo J, Sokal E, Kieninger D, Prymula R, Dull PM, Kohl I, Barone M, Wang H, Toneatto D, Pollard AJ; European MenB Vaccine Study Group. Persistence of Bactericidal Antibodies After Infant Serogroup B Meningococcal Immunization and Booster Dose Response at 12, 18 or 24 Months of Age. Pediatr Infect Dis J. 2016 Apr;35(4):e113-23. doi: 10.1097/INF.0000000000001056. PMID 26756390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 6 centres in Belgium, 4 in Czech, 24 in Germany, 5 in Italy, 16 in Spain and 4 in UK who had previously participated in and completed the study V72P12.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- B+R246_12: Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age.age
Period: Overall Study
Arm/Group | B+R246_12 | B+R246_18 | B+R246_24 | B246_12 | B246_18 | B246_24 | B+R234_12 | B+R234_18 | B+R234_24 | B12 14 | B18 20 | B24 26
Started | 188 | 157 | 152 | 174 | 164 | 143 | 106 | 78 | 73 | 246 | 51 | 56
Completed | 183 | 150 | 143 | 170 | 150 | 123 | 102 | 73 | 63 | 236 | 50 | 52
Not Completed | 5 | 7 | 9 | 4 | 14 | 20 | 4 | 5 | 10 | 10 | 1 | 4
Not completed — Inappropriate enrollment | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 6 | 2 | 5 | 8 | 2 | 2 | 3 | 4 | 0 | 4
Not completed — Lost to Follow-up | 0 | 4 | 2 | 0 | 5 | 7 | 0 | 1 | 5 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 1 | 2 | 3 | 0 | 1 | 1 | 4 | 0 | 0
Not completed — Unable to classify | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Administrative reason | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B+R246_12 | B+R246_18 | B+R246_24 | B246_12 | B246_18 | B246_24 | B+R234_12 | B+R234_18 | B+R234_24 | B12 14 | B18 20 | B24 26 | Total
Number analyzed (Participants) | 188 | 157 | 152 | 174 | 164 | 143 | 106 | 78 | 73 | 246 | 51 | 56 | 1588
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 188 | 157 | 152 | 174 | 164 | 143 | 106 | 78 | 73 | 246 | 51 | 56 | 1588
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.6 (1.2) | 18.1 (0.6) | 24 (0.4) | 12.7 (0.9) | 18.1 (0.5) | 24 (0.3) | 12.8 (1.4) | 18 (0.4) | 24 (0.5) | 12.6 (1.3) | 18 (0.2) | 24 (0.2) | 17.1 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 73 | 77 | 81 | 80 | 75 | 62 | 41 | 34 | 115 | 23 | 23 | 762
  Male | 110 | 84 | 75 | 93 | 84 | 68 | 44 | 37 | 39 | 131 | 28 | 33 | 826

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Serum Bactericidal Antibody Titers ≥1:5 After Receiving a Fourth (Booster) Dose of rMenB+OMV NZ Vaccination in Subjects Who Previously Received 3 Doses of rMenB+OMV NZ and Routine Vaccines at 2, 4 and 6 Months of Age.
Description: Immunogenicity was assessed in terms of percentage of subjects with serum bactericidal antibody (SBA) titers ≥1:5 (98.3% CI) against N.meningitidis serogroup reference strains H44/76, NZ98/254 and 5/99, one month after the fourth (booster) dose of meningococcal B vaccine at 12 or 18 or24 months of age who were previously vaccinated with 3 doses of rMenB+OMV NZ and routine vaccines at 2, 4 and 6 months of age.
Time Frame: 1 month after booster
Population: The analysis was performed on the per-protocol population. This outcome measure was assessed only for the strains H44/76, NZ98/254 and 5/99. As exploratory analyses were performed on the M10713 strain, no endpoints were considered for this strain.
Measure: Number (98.3% Confidence Interval); unit: percentage of subjects
Arm/Group | B+R246_12 | B+R246_18 | B+R246_24
Number analyzed (Participants) | 162 | 120 | 108
percentage of subjects
  hSBA≥ 1: 5 (H44/76 strain)(N = 158,116,101) | 97 [93 to 99] | 100 [96 to 100] | 100 [95 to 100]
  hSBA≥ 1: 5 (5/99 strain)(N= 156,118,100) | 100 [97 to 100] | 100 [96 to 100] | 100 [95 to 100]
  hSBA≥ 1: 5 (NZ 98/254 strain)(N= 159,118,103) | 95 [89 to 98] | 77 [67 to 86] | 84 [74 to 92]
  hSBA≥ 1: 5 (M10713 strain) | NA [NA to NA] — In this group exploratory analyses was not performed | NA [NA to NA] — In this group exploratory analyses was not performed | NA [NA to NA] — In this group exploratory analyses was not performed

2. Secondary Outcome: Percentages of Subjects With SBA Titers ≥1:5 After Receiving a Fourth (Booster) Dose of rMenB+OMV NZ Vaccination in Subjects Who Previously Received 3 Doses of rMenB+OMV NZ at 2, 4 and 6 Months of Age and Routine Vaccines at 3, 5 and 7 Months of Age.
Description: Immunogenicity was assessed in terms of Percentages of Subjects With SBA Titers ≥1:5 (98.3% CI), After Receiving a Fourth (Booster) Dose of rMenB+OMV NZ Vaccination in subjects who previously received 3 doses of rMenB+OMV NZ at 2, 4 and 6 months of age and routine vaccines at 3, 5 and 7 months of age.
Time Frame: 1 month after booster
Population: The analysis was performed on per-protocol population. This outcome measure was assessed only against H44/76, NZ98/254 and 5/99 strains. As exploratory analyses were performed on the M10713 strain, no endpoints were considered for this strain.
Measure: Number (98.3% Confidence Interval); unit: percentage of subjects
Arm/Group | B246_12 | B246_18 | B246_24
Number analyzed (Participants) | 145 | 114 | 98
percentage of subjects
  hSBA≥ 1: 5 (H44/76 strain)(N= 138,111,93) | 100 [97 to 100] | 99 [94 to 100] | 100 [95 to 100]
  hSBA≥ 1: 5 (5/99 strain)(N= 142,110,92) | 100 [97 to 100] | 100 [96 to 100] | 100 [95 to 100]
  hSBA≥ 1: 5 (NZ 98/254 strain)(N= 142,111,95) | 96 [90 to 99] | 86 [76 to 93] | 89 [80 to 96]
  hSBA≥ 1: 5 (M10713 strain) | NA [NA to NA] — In this group exploratory analyses was not performed | NA [NA to NA] — In this group exploratory analyses was not performed | NA [NA to NA] — In this group exploratory analyses was not performed

3. Secondary Outcome: Percentages of Subjects With Serum Bactericidal Antibody Titers ≥1:5 After Receiving a Fourth (Booster) Dose of rMenB+OMV NZ Vaccination in Subjects Who Previously Received 3 Doses of rMenB+OMV NZ and Routine Vaccines at 2, 3 and 4 Months of Age.
Description: Immunogenicity was assessed in terms of percentage of subjects with serum bactericidal antibody (SBA) titers ≥1:5 (98.3% CI) against N.meningitidis serogroup reference strains H44/76, NZ98/254 and 5/99, one month after the fourth (booster) dose of meningococcal B vaccine at 12 or 18 or24 months of age who were previously vaccinated with 3 doses of rMenB+OMV NZ and routine vaccines at 2, 3 and 4 months of age.
Time Frame: 1 month after booster
Population: The analysis was performed on the per-protocol population
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | B+R234_12 | B+R234_18 | B+R234_24
Number analyzed (Participants) | 86 | 58 | 48
percentage of subjects
  hSBA≥ 1: 5 (H44/76 strain)(N= 83,56,48 ) | 100 [94 to 100] | 98 [88 to 100] | 100 [91 to 100]
  hSBA≥ 1: 5 (5/99 strain)(N= 84,56,46) | 100 [94 to 100] | 100 [92 to 100] | 100 [90 to 100]
  hSBA≥ 1: 5 (NZ 98/254 strain)(N= 83,56,48) | 97 [89 to 100] | 80 [65 to 91] | 96 [83 to 100]
  hSBA≥ 1: 5 (M10713 strain)(N= 67,50,41) | 76 [62 to 87] | 74 [57 to 87] | 95 [81 to 100]

4. Secondary Outcome: Geometric Mean Titers (GMTs) in Subjects One Month After Receiving a Fourth (Booster) Dose of rMenB+OMV NZ Vaccination in Subjects at 12 18 or 24 Months of Age Who Previously Received 3 Doses of rMenB+OMV NZ at 2, 3 and 4 or 2, 4 and 6 Months of Age.
Description: The serum antibody titers one month after the fourth (booster) dose of meningococcal B vaccine at 12 or 18 or24 months of age who were previously vaccinated with 3 doses of rMenB+OMV NZ at 2, 3 and 4 or 2, 4 and 6 months of age, are reported as geometric mean titers (GMTs) against N.meningitidis serogroup reference strains H44/76, NZ98/254 and 5/99.
Time Frame: 1 month after booster
Population: The analysis was performed on the per-protocol population. For hSBA≥ 1: 5 (H44/76 strain) (N=158 116 101 138 111 93 83 56 48) For hSBA≥ 1: 5 (5/99 strain) (N=156 118 100 142 110 92 84 56 46) For hSBA≥ 1: 5 (NZ 98/254 strain) (N=159 118 103 142 111 95 86 56 48) For hSBA≥ 1: 5 (M10713 strain) (N=0 0 0 0 0 0 67 50 41)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+R246_12 | B+R246_18 | B+R246_24 | B246_12 | B246_18 | B246_24 | B+R234_12 | B+R234_18 | B+R234_24
Number analyzed (Participants) | 162 | 120 | 108 | 145 | 114 | 98 | 86 | 58 | 48
Titers
  hSBA≥ 1: 5 (H44/76 strain) | 125 [106 to 148] | 123 [101 to 149] | 108 [88 to 133] | 178 [149 to 213] | 164 [135 to 200] | 152 [122 to 188] | 135 [108 to 170] | 92 [70 to 121] | 128 [95 to 172]
  hSBA≥ 1: 5 (5/99 strain) | 1276 [1092 to 1491] | 2183 [1824 to 2611] | 1820 [1497 to 2212] | 1713 [1454 to 2020] | 2058 [1710 to 2476] | 2739 [2233 to 3361] | 1558 [1262 to 1923] | 1486 [1148 to 1924] | 2081 [1564 to 2771]
  hSBA≥ 1: 5 (NZ 98/254 strain) | 36 [29 to 44] | 15 [12 to 19] | 17 [14 to 22] | 34 [27 to 42] | 17 [14 to 22] | 19 [15 to 25] | 47 [36 to 62] | 17 [12 to 24] | 33 [23 to 47]
  hSBA≥ 1: 5 (M10713 strain) | NA [NA to NA] — In this group exploratory analyses was not performed. | NA [NA to NA] — In this group exploratory analyses was not performed. | NA [NA to NA] — In this group exploratory analyses was not performed. | NA [NA to NA] — In this group exploratory analyses was not performed. | NA [NA to NA] — In this group exploratory analyses was not performed. | NA [NA to NA] — In this group exploratory analyses was not performed. | 12 [8.52 to 17] | 15 [10 to 23] | 26 [17 to 41]

5. Secondary Outcome: GMTs in Subjects One Month After the Fourth (Booster) Dose of Meningococcal B Vaccine at 12 Months of Age Previously Vaccinated With 3 Doses of rMenB+OMV NZ at 2, 3 and 4 or 2, 4 and 6 Months of Age and Single Dose of rMenB+OMV NZ Given at Same Age
Description: Characterization of immunological memory by serum antibody titers (98.3% CI) one month after the fourth (booster) dose of meningococcal B vaccine at 12 months of age who were previously vaccinated with 3 doses of rMenB+OMV NZ at 2, 3 and 4 or 2, 4 and 6 months of age and single dose of rMenB+OMV NZ given at same ages, are reported as geometric mean titers (GMTs) against N.meningitidis serogroup reference strains H44/76, NZ98/254 and 5/99.
Time Frame: 1 month after booster
Population: The analysis was performed on the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+R246_12 | B246_12 | B+R234_12 | B12 14
Number analyzed (Participants) | 162 | 145 | 86 | 239
Titers
  hSBA≥ 1: 5 (H44/76 strain)(N= 158,138,83,217) | 125 [102 to 154] | 179 [144 to 223] | 137 [104 to 181] | 18 [15 to 21]
  hSBA≥ 1: 5 (5/99 strain)(N= 156,142,84,216) | 1301 [1076 to 1573] | 1763 [1441 to 2157] | 1607 [1243 to 2077] | 49 [42 to 58]
  hSBA≥ 1: 5 (NZ 98/254 strain)(N= 159,142,86,220) | 37 [29 to 46] | 35 [27 to 44] | 48 [36 to 65] | 3.71 [3.06 to 4.5]

6. Secondary Outcome: GMTs in Subjects One Month After the Fourth (Booster) Dose of Meningococcal B Vaccine at 18 and 24months of Age, Previously Vaccinated With 3 Doses of rMenB+OMV NZ at 2, 3 and 4 or 2, 4 and 6 Months of Age and Single Dose of rMenB+OMV NZ Given at Same Age
Description: Characterization of immunological memory by serum antibody titers one month after the fourth (booster) dose of meningococcal B vaccine at 18 and 24months of age who were previously vaccinated with 3 doses of rMenB+OMV NZ at 2, 3 and 4 or 2, 4 and 6 months of age and single dose of rMenB+OMV NZ given at same ages, are reported as geometric mean titers (GMTs) against N.meningitidis serogroup reference strains H44/76, NZ98/254 and 5/99.
Time Frame: 1 month after booster
Population: The analysis was performed on the per-protocol population. For hSBA≥ 1: 5 (H44/76 strain)(N=116 101 111 93 56 48 46 52), hSBA≥ 1: 5 (5/99 strain) (N=118 100 110 92 56 46 48 50), hSBA≥ 1: 5 (NZ 98/254 strain) (N=118 103 111 95 56 48 47 50)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+R246_18 | B+R246_24 | B246_18 | B246_24 | B+R234_18 | B+R234_24 | B18 20 | B24 26
Number analyzed (Participants) | 120 | 108 | 114 | 98 | 58 | 48 | 47 | 53
Titers
  hSBA≥ 1: 5 (H44/76 strain) | 126 [104 to 154] | 110 [89 to 136] | 162 [132 to 198] | 155 [124 to 193] | 93 [70 to 123] | 132 [97 to 180] | 18 [13 to 25] | 14 [10 to 19]
  hSBA≥ 1: 5 (5/99 strain) | 2195 [1790 to 2691] | 1811 [1449 to 2262] | 2034 [1648 to 2511] | 2735 [2166 to 3455] | 1483 [1107 to 1986] | 2087 [1508 to 2889] | 41 [30 to 56] | 30 [22 to 41]
  hSBA≥ 1: 5 (NZ 98/254 strain) | 16 [12 to 20] | 18 [14 to 23] | 17 [14 to 22] | 20 [15 to 26] | 17 [12 to 25] | 34 [23 to 49] | 2.76 [1.87 to 4.08] | 2.1 [1.44 to 3.07]

7. Secondary Outcome: Two-dose Catch-up Regimen of rMenB+OMV NZ in Unprimed Toddlers Aged 12, 18 or 24 Months
Description: Immunogenicity evaluation of a two-dose catch-up regimen of rMenB+OMV NZ in unprimed toddlers aged 12, 18 or 24 months as measured by serum antibody titers one month after the second vaccination f meningococcal B vaccine at 18 and 24months of age who were previously vaccinated with 3 doses of rMenB+OMV NZ reported as geometric mean titers (GMTs) against N.meningitidis serogroup reference strains H44/76, NZ98/254 and 5/99.
Time Frame: 1 month after second vaccination
Population: The analysis was performed on the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B12 14 | B18 20 | B24 26
Number analyzed (Participants) | 189 | 44 | 49
Titers
  hSBA≥ 1: 5 (H44/76 strain)(N= 156,42,45) | 188 [164 to 216] | 171 [130 to 224] | 177 [136 to 231]
  hSBA≥ 1: 5 (5/99 strain)(N= 177, 40,46) | 635 [548 to 735] | 491 [359 to 672] | 559 [417 to 749]
  hSBA≥ 1: 5 (NZ 98/254 strain)(N = 179,44,45) | 40 [35 to 47] | 23 [17 to 30] | 24 [18 to 32]
  hSBA≥ 1: 5 (M10713 strain)(N= 0,34,37) | NA [NA to NA] — In this group exploratory analyses was not performed. | 14 [8.02 to 23] | 18 [11 to 29]

8. Secondary Outcome: Geometric Mean Concentrations Against Vaccine Antigen 287- 953 One Month After Fourth Booster Dose to Previously Primed Toddlers at 12, 18 or 24 Months of Age.
Description: Immunogenicity evaluation against vaccine antigen 287-953 one month after fourth booster dose to previously primed toddlers at 12, 18 or 24 months measured by ELISA.
Time Frame: 1 month after booster vaccination
Population: The analysis was performed on the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | B+R246_12 | B+R246_18 | B+R246_24 | B246_12 | B246_18 | B246_24 | B+R234_12 | B+R234_18 | B+R234_24
Number analyzed (Participants) | 162 | 119 | 108 | 145 | 114 | 98 | 86 | 58 | 48
IU/mL | 5334 [4670 to 6093] | 6395 [5474 to 7470] | 6864 [5826 to 8087] | 6605 [5733 to 7609] | 6418 [5477 to 7520] | 8120 [6833 to 9649] | 6125 [5110 to 7342] | 5952 [4771 to 7426] | 6774 [5305 to 8649]

9. Secondary Outcome: Geometric Mean Concentrations Against Vaccine Antigen 287- 953 One Month After Booster Given After a Two-dose Catch-up Regimen in Toddlers Starting at 12, 18 or 24 Months of Age.
Description: Immunogenicity evaluation against vaccine antigen 287-953 one month after booster given after a two-dose catch-up regimen in toddlers starting at 12, 18 or 24 months of age.one month after fourth booster dose to previously primed toddlers at 12, 18 or 24 months of age measured by ELISA
Time Frame: 1 month after booster vaccination
Population: The analysis was performed on the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | B12 14 | B18 20 | B24 26
Number analyzed (Participants) | 177 | 44 | 47
IU/mL | 122 [101 to 147] | 121 [84 to 176] | 100 [69 to 144]

10. Secondary Outcome: Number of Children Reporting Solicited Local and Systemic Adverse Events After Receiving a Fourth Booster Dose of rMenB+OMV NZ Vaccine at 12, 18 or 24 Months of Age.
Description: The safety and tolerability of the 4th booster dose rMenB+OMV NZ vaccine in children (12, 18 or 24 months age) is reported as number of subjects with solicited local and systemic adverse events.
Time Frame: From day 1 to day 7 after vaccination
Population: Analysis was done on the Safety Population.
Measure: Number; unit: participants
Arm/Group | B246_12 | B246_18 | B246_24
Number analyzed (Participants) | 170 | 153 | 126
participants
  Any | 156 | 135 | 116
  Any Local | 137 | 119 | 113
  Injection site Tenderness | 104 | 104 | 105
  Injection site Erythema | 117 | 94 | 94
  Injection site Induration | 93 | 62 | 73
  Injection site Swelling | 57 | 52 | 50
  Any Systemic | 134 | 118 | 101
  ChangeEat.Habits | 66 | 59 | 51
  Sleepiness | 63 | 56 | 52
  Vomiting | 8 | 9 | 8
  Diarrhea | 37 | 23 | 27
  Irritbility | 104 | 91 | 83
  Unusual Crying | 52 | 51 | 40
  Rash | 7 | 3 | 7
  Fever ( >= 38C ) | 52 | 55 | 28
  Any Ohter | 59 | 59 | 40
  Body Temp. <38 C | 118 | 98 | 98
  Medical Attend. Fever | 5 | 5 | 2
  Antipyretic prophylactic | 32 | 28 | 25
  Antipyretic therapeutic | 37 | 39 | 21

11. Secondary Outcome: Number of Children Reporting Solicited Local and Systemic Adverse Events After Receiving a Two-dose Catch-up Regimen of rMenB+OMV NZ Vaccine at 12, 18 or 24 Months of Age.
Description: The safety and tolerability of the two-dose catch-up regimen of rMenB+OMV NZ vaccine in children (12, 18 or 24 months age) is reported as number of subjects with solicited local and systemic adverse events.
Time Frame: day 1 to day 7 after vaccination
Population: The analysis was done on safety population
Measure: Number; unit: participants
Arm/Group | B12 14 | B18 20 | B24 26
Number analyzed (Participants) | 239 | 51 | 55
participants
  Injection site Tenderness (vaccination 1) | 151 | 35 | 47
  Injection site Tenderness (vaccination 2) | 143 | 32 | 42
  Injection site Erythema (vaccination 1) | 151 | 32 | 39
  Injection site Erythema (vaccination 2) | 148 | 33 | 31
  Injection site Induration (vaccination 1) | 112 | 20 | 27
  Injection site Induration (vaccination 2) | 101 | 24 | 22
  Injection site Swelling (vaccination 1) | 81 | 15 | 19
  Injection site Swelling (vaccination 2) | 72 | 18 | 19
  Change in Eating habits (vaccination 1) | 95 | 13 | 25
  Change in Eating habits (vaccination 2) | 83 | 19 | 21
  Sleepiness (vaccination 1) | 106 | 21 | 18
  Sleepiness (vaccination 2) | 78 | 16 | 18
  Vomiting (vaccination 1) | 19 | 5 | 6
  Vomiting (vaccination 2) | 18 | 1 | 4
  Diarrhea (vaccination 1) | 43 | 13 | 20
  Diarrhea (vaccination 2) | 35 | 5 | 7
  Irritability (vaccination 1) | 156 | 23 | 28
  Irritability (vaccination 2) | 126 | 27 | 23
  Unusual Crying (vaccination 1) | 81 | 13 | 15
  Unusual Crying (vaccination 2) | 67 | 14 | 15
  Rash (vaccination 1) | 13 | 5 | 2
  Rash (vaccination 2) | 10 | 4 | 0
  Fever ( >= 38C ) (vaccination 1) | 83 | 14 | 15
  Fever ( >= 38C ) (vaccination 2) | 74 | 15 | 13
  Body Temp.<38 C (vaccination 1) | 156 | 37 | 39
  Body Temp.<38 C (vaccination 2) | 163 | 36 | 39
  Medical Attend. Fever (vaccination 1) | 9 | 2 | 1
  Medical Attend. Fever (vaccination 2) | 5 | 1 | 0
  Antipyretic prophylactic (vaccination 1) | 49 | 8 | 8
  Antipyretic prophylactic (vaccination 2) | 45 | 9 | 11
  Antipyretic therapeutic (vaccination 1) | 66 | 9 | 11
  Antipyretic therapeutic (vaccination 2) | 54 | 11 | 7

ADVERSE EVENTS:
Time Frame: From day 1 to day 7 after vaccination
Description: Of the 1588 subjects enrolled into this study, 1519 were vaccinated and included in the safety analysis.
Arm/Group | B+R246_12 | B+R246_18 | B+R246_24 | B246_12 | B246_18 | B246_24 | B+R234_12 | B+R234_18 | B+R234_24 | B12 14 | B18 20 | B24 26
Serious Adverse Events (participants affected / at risk) | 5/185 | 3/152 | 6/144 | 6/170 | 7/153 | 1/126 | 5/104 | 5/74 | 3/66 | 16/239 | 0/51 | 1/55
Other Adverse Events (participants affected / at risk) | 180/185 | 147/152 | 140/144 | 163/170 | 139/153 | 116/126 | 102/104 | 73/74 | 62/66 | 230/239 | 50/51 | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B+R246_12 (N=185) | B+R246_18 (N=152) | B+R246_24 (N=144) | B246_12 (N=170) | B246_18 (N=153) | B246_24 (N=126) | B+R234_12 (N=104) | B+R234_18 (N=74) | B+R234_24 (N=66) | B12 14 (N=239) | B18 20 (N=51) | B24 26 (N=55)
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petit mal Epilepsy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Congenital aural fistula (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Walking disability (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coeliac Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acetonaemic vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Gastroenteritis Rotavirus (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema herpeticum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Superinfection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B+R246_12 (N=185) | B+R246_18 (N=152) | B+R246_24 (N=144) | B246_12 (N=170) | B246_18 (N=153) | B246_24 (N=126) | B+R234_12 (N=104) | B+R234_18 (N=74) | B+R234_24 (N=66) | B12 14 (N=239) | B18 20 (N=51) | B24 26 (N=55)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 12 | 5 | 13 | 8 | 7 | 3 | 4 | 2 | 24 | 6 | 8
Somnolence (Nervous system disorders) | 72 | 61 | 72 | 63 | 56 | 52 | 50 | 33 | 27 | 129 | 25 | 28
Crying (General disorders) | 56 | 43 | 46 | 52 | 51 | 40 | 41 | 18 | 22 | 105 | 17 | 25
Induration (General disorders) | 2 | 0 | 2 | 3 | 3 | 4 | 2 | 0 | 0 | 2 | 1 | 4
Injection site erythema (General disorders) | 127 | 100 | 109 | 117 | 94 | 94 | 76 | 52 | 49 | 179 | 38 | 41
Injection site induration (General disorders) | 101 | 74 | 76 | 93 | 62 | 73 | 52 | 41 | 35 | 148 | 27 | 33
Injection site pain (General disorders) | 107 | 114 | 118 | 104 | 104 | 105 | 70 | 56 | 51 | 187 | 41 | 51
Injection site swelling (General disorders) | 73 | 53 | 63 | 57 | 52 | 50 | 32 | 36 | 25 | 107 | 21 | 24
Pyrexia (General disorders) | 78 | 57 | 50 | 60 | 59 | 32 | 53 | 28 | 27 | 133 | 24 | 22
Swelling (General disorders) | 1 | 1 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 3
Eating disorder (Psychiatric disorders) | 64 | 70 | 68 | 66 | 59 | 51 | 41 | 29 | 28 | 126 | 21 | 34
Irritability (Psychiatric disorders) | 110 | 100 | 92 | 104 | 91 | 83 | 72 | 53 | 44 | 177 | 32 | 35
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 39 | 26 | 32 | 40 | 27 | 27 | 21 | 18 | 13 | 72 | 16 | 21
Enteritis (Gastrointestinal disorders) | 5 | 0 | 1 | 2 | 3 | 3 | 2 | 1 | 2 | 4 | 3 | 1
Teething (Gastrointestinal disorders) | 8 | 3 | 1 | 2 | 0 | 0 | 3 | 2 | 0 | 15 | 1 | 0
Vomiting (Gastrointestinal disorders) | 15 | 16 | 11 | 13 | 12 | 10 | 15 | 8 | 2 | 41 | 7 | 8
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 9 | 2 | 2 | 6 | 5 | 0 | 2 | 4 | 0 | 13 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 2 | 2 | 1 | 0 | 1 | 3 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 9 | 9 | 20 | 8 | 5 | 9 | 10 | 7 | 5 | 26 | 8 | 4
Bronchitis (Infections and infestations) | 7 | 11 | 5 | 19 | 7 | 5 | 9 | 6 | 4 | 19 | 3 | 9
Candida nappy rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 3 | 1
Conjunctivitis (Infections and infestations) | 11 | 11 | 3 | 10 | 10 | 7 | 5 | 1 | 3 | 15 | 4 | 4
Ear infection (Infections and infestations) | 12 | 8 | 6 | 13 | 5 | 6 | 14 | 5 | 3 | 29 | 6 | 4
Fungal infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
Gastroenteritis (Infections and infestations) | 17 | 6 | 4 | 9 | 5 | 7 | 4 | 2 | 0 | 10 | 4 | 2
Infection (Infections and infestations) | 1 | 0 | 2 | 0 | 3 | 2 | 2 | 1 | 1 | 2 | 3 | 3
Influenza (Infections and infestations) | 3 | 4 | 1 | 3 | 2 | 1 | 0 | 2 | 0 | 1 | 1 | 5
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 20 | 6 | 12 | 13 | 12 | 4 | 7 | 5 | 2 | 21 | 8 | 7
Otitis media (Infections and infestations) | 3 | 6 | 2 | 6 | 4 | 2 | 3 | 2 | 4 | 11 | 2 | 4
Pharyngitis (Infections and infestations) | 7 | 8 | 3 | 5 | 14 | 6 | 5 | 3 | 3 | 16 | 3 | 1
Respiratory tract infection (Infections and infestations) | 9 | 3 | 2 | 6 | 3 | 3 | 5 | 2 | 2 | 8 | 5 | 6
Rhinitis (Infections and infestations) | 10 | 5 | 4 | 12 | 4 | 7 | 4 | 3 | 1 | 17 | 2 | 5
Scarlet fever (Infections and infestations) | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Tonsillitis (Infections and infestations) | 6 | 9 | 7 | 9 | 6 | 3 | 5 | 3 | 3 | 14 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 10 | 8 | 0 | 6 | 15 | 5 | 10 | 2 | 0 | 18 | 2 | 5
Varicella (Infections and infestations) | 4 | 1 | 2 | 2 | 2 | 7 | 2 | 0 | 5 | 9 | 5 | 1
Viral infection (Infections and infestations) | 12 | 6 | 6 | 7 | 10 | 5 | 5 | 5 | 6 | 21 | 8 | 3

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.